CLINICAL TRIAL: NCT00113061
Title: INFLAME: Inflammation and Exercise
Brief Title: Effect of Exercise on Elevated C-reactive Protein Concentrations in Formerly Inactive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 180; R01HL075442 (NIH)
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2007-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
Keywords: Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity | interventions — Exercise

INTERVENTIONS:
Procedure: Exercise

SUMMARY:
The purpose of this study is to determine the effect of exercise training on elevated C-reactive protein (CRP) concentrations, an indicator of inflammation, in initially inactive women and men.

DETAILED DESCRIPTION:
BACKGROUND:

CRP, a marker of systemic inflammation, has been reported to be an independent predictor of cardiovascular disease in both women and men. Recently published data from cross-sectional analyses showed that CRP is inversely related to cardiorespiratory fitness, and that this association is independent of body mass index. Regular exercise may affect CRP levels, and can possibly be used as a means of reducing elevated CRP levels. Though there are a number of studies focusing on related topics, there are no published reports from randomized clinical trials on the effect of exercise training alone on CRP levels.

DESIGN NARRATIVE:

An estimated 200 individuals will be randomly assigned to either a no exercise control group or an exercise group. Exercising individuals will participate in 3 or 4 training sessions each week for 4 months, and will progress to a total energy expenditure of 16 kcal [kg(-1), week(-1)], which is an exercise dose at the upper end of current public health recommendations for physical activity. The target exercise intensity will be 50-70% of baseline volume of oxygen consumed (V02 max). VO2 max is the maximal rate of oxygen consumption during exercise, and is a measurement of fitness. The primary outcome measure will be plasma CRP concentration. Secondary outcomes will be changes in variables that are potential mechanisms through which regular exercise might reduce CRP. These variables include visceral adiposity, the cytokines interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha), and heart rate variability as a measure of autonomic balance. Although the primary outcome is CRP level, this study will also contribute significantly to the limited body of literature examining the effect of exercise on the variables of visceral adiposity, cytokines, and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive
* C-reactive protein level at least 2.0 mg/L but less than 10.0 mg/L upon study entry
* Body mass index between 18.5 kg/square meter and 40.0 kg/square meter as measured at study entry
* Does not smoke
* Total cholesterol at least 240 mg/dl with LDL-C at least 160 mg/dl OR LDL less than 190 mg/dl and Framingham less than 10%
* Triglyceride levels no higher than 300 mg/dl
* Fasting glucose level less than 126
* Systolic blood pressure less than 140 mm Hg and/or diastolic blood pressure less than 90 mm Hg as measured at study entry
* If taking an oral contraceptive, aspirin, ibuprofen, or other anti-inflammatory medications, must be on a stable dose for 6 months prior to study entry
* If taking a cholesterol medication, including statins, blood pressure medication (including ace inhibitors), or multi-vitamins, must be on a stable dose for 2 months prior to study entry

Exclusion Criteria:

* Using a beta blocker, hormone replacement therapy, or corticosteroids (except inhalers)
* Any rheumatologic, orthopedic, neurological, or autoimmune diseases, or seizure disorder
* Any significant cardiovascular disease or disorders including, but not limited to, stent or coronary artery bypass grafting
* Cardiac dysrhythmias including, but not limited to, left bundle branch block, atrial fibrillation, pacemaker, or automatic implantable cardioverter defibrillator
* Any surgery, broken bones, blood donation, or anaphylactic shock within 6 months of study entry
* Any sprain or strain, removal of wisdom teeth, or use of antibiotics within 3 months of study entry
* History of stroke or TIA
* History of cancer within at least 5 years of study entry
* Diabetes or glucose intolerance
* Planning on participating in any other research trials during the next year
* Currently pregnant
* Planning to becoming pregnant during the next year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162
Dates: Start 2004-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Plasma CRP concentration (measured at Month 4)

SECONDARY OUTCOMES:
Changes in visceral adiposity, the cytokines interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha), and heart rate variability (measured at Month 4)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S. Church, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, LSU System, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Church TS, Earnest CP, Thompson AM, Priest EL, Rodarte RQ, Saunders T, Ross R, Blair SN. Exercise without weight loss does not reduce C-reactive protein: the INFLAME study. Med Sci Sports Exerc. 2010 Apr;42(4):708-16. doi: 10.1249/MSS.0b013e3181c03a43. PMID 19952828